CLINICAL TRIAL: NCT04738396
Title: Electrogram and Hemodynamic Characteristics of Adaptive LBBAP in Patients With Heart Failure or Bradycardia
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: aLBBAP study
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Cardiac Pacing; Pacing Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-site, non-randomized, data collection study. The purpose of this study is to investigate the cardiac electrical and mechanical function during LBBAP with different AV intervals.

DETAILED DESCRIPTION:
Left bundle branch pacing (LBBP), achieved via trans-septal approach with the pacing tip at the left side of the ventricular septum, has recently initiated and been well practiced in China. LBBP is characterized with relatively ease of implantation (usually <5 minutes fluoroscopic use time), narrow paced QRS duration (similar to physiological pacing), low and stable pacing threshold (usually around 0.5V @0.5ms, good for device longevity and long-term stability without need of back-up pacing lead), high R wave amplitude for pacing management, and LBBB (left bundle branch block) correction by a low pacing output.

LBBAP (left bundle branch area pacing) can generate a relatively narrow QRSd and fast left ventricular activation. As AV interval is an important pacing parameter relevant to cardiac function. This study is to investigate the cardiac electrical and mechanical function during LBBAP with different AV intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 80 years old
* Patients who are willing to provide Informed Consent
* Patients who received LBBAP for at least 3 months
* Patients' implanted device can provide intracardiac electrograms
* Bradycardia patients with AVB or heart failure patients with LBBB

Exclusion Criteria:

* Patients who are pregnant or have a plan for pregnancy during the study
* Patients with persistent AF
* Patients who have medical conditions that would limit study participation
* Patients who were already enrolled in other clinical trial which would impact his/her participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received LBBAP for at least 3 months and come back to hospital for regular follow-up will be considered to be recruited voluntarily.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
ECG QRS duration | At least 3 months post implant
  The primary endpoint is QRS duration during LBBP

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong Zhou, Study Director — Medtronic
Locations (4):
- China (4):
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Greentown Cardiovascular Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang